CLINICAL TRIAL: NCT01825226
Title: THE IMPACT OF THE ENHANCED HOMESTEAD FOOD PRODUCTION PROGRAM ON CHILD HEALTH
Brief Title: Helen Keller International's Enhanced-Homestead Food Production Program in Burkina Faso
Acronym: EHFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6117001
Record Dates: First submitted 2013-01-01; First posted 2013-04-05 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Growth; Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Program participation (Experimental): Participation in an enhanced-homestead food production program including home gardening and nutrition and health behavior change communication
  Interventions: Other: Enhanced-Homestead Food Production Program
- Control (No Intervention)

INTERVENTIONS:
Other: Enhanced-Homestead Food Production Program — Participation in an enhanced-homestead food production program including home gardening and nutrition and health behavior change communication
  Arms: Program participation

SUMMARY:
Helen Keller International (HKI) has been implementing homestead food production (HFP) programs in Asia for the past 20 years and has recently begun implementing HFP programs in Africa as well. In general, these programs target women and are designed to improve maternal and child health and nutrition outcomes through three primary pathways: 1. Increasing the availability of micronutrient-rich foods through increased household production of these foods; 2. Raising income through the sale of surplus production; and 3. Increasing knowledge and adoption of optimal nutrition practices, including the consumption of micronutrient-rich foods. Evaluations of HFP programs have consistently demonstrated significant increases in household production and consumption of micronutrient-rich foods. This increased consumption, along with improvements in health and nutrition related knowledge, and increased income, could all contribute to improvements in maternal and child health and nutrition outcomes. However, to date there has been limited understanding as to how these types of programs can be optimized to maximize impacts on these outcomes.

In order to better understand the potential of these types of programs to improve maternal and child health and nutrition outcomes and how this impact may be achieved IFPRI has been collaborating with HKI to evaluate one of their E-HFP programs in Burkina Faso. The evaluation considers impact of the program through the three pathways above, and assesses anthropometric and clinical measures of nutrition, as well as looking at how the programs might be improved.

ELIGIBILITY:
Inclusion Criteria:

* Mother of child between the ages of 3 and 12 months and her child

Exclusion Criteria:

* N/A

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1763 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
Growth | Measurements will be made for children between the ages of 3 and 12 months of age at baseline and then 2 years later, at endline, when the children are between the ages of 23 and 40 months
  Change in height-for-age Z-scores, weight-for-age Z-scores and weight-for-height Z-scores will be measured as well as the change in the prevalence of stunting (HAZ <-2), underweight (WAZ <-2) and wasting (WHZ <-2) over the course of the two year program period.
Hemoglobin | Measurements will be made for children between the ages of 3 and 12 months of age at baseline and then 2 years later, at endline, when the children are between the ages of 23 and 40 months

SECONDARY OUTCOMES:
Food security | Baseline (2010), Endline (2012), follow-up (2013)
Household assets | Baseline (2010), Endline (2012), follow-up (2013)
Household consumption | Baseline (2010), Endline (2012), follow-up (2013)
Household livestock holdings | Baseline (2010), Endline (2012), follow-up (2013)
Dietary diversity | Baseline (2010), Endline (2012), follow-up (2013)
Mother's BMI | Baseline (2010), Endline (2012), follow-up (2013)
Maternal health and nutrition-related knowledge | Baseline (2010), Endline (2012), follow-up (2013)
IYCF practices | Baseline (2010), Endline (2012), follow-up (2013)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna K Olney, Ph.D., Principal Investigator — International Food Policy Research Institute; Andrew Dillon, Ph.D., Principal Investigator — Michigan Sate University
Locations (1):
- International Food Policy Research Institute, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Nielsen JN, Olney DK, Ouedraogo M, Pedehombga A, Rouamba H, Yago-Wienne F. Process evaluation improves delivery of a nutrition-sensitive agriculture programme in Burkina Faso. Matern Child Nutr. 2018 Jul;14(3):e12573. doi: 10.1111/mcn.12573. Epub 2017 Dec 26. PMID 29278449
- [Derived] Olney DK, Bliznashka L, Pedehombga A, Dillon A, Ruel MT, Heckert J. A 2-Year Integrated Agriculture and Nutrition Program Targeted to Mothers of Young Children in Burkina Faso Reduces Underweight among Mothers and Increases Their Empowerment: A Cluster-Randomized Controlled Trial. J Nutr. 2016 May;146(5):1109-17. doi: 10.3945/jn.115.224261. Epub 2016 Apr 13. PMID 27075910
- [Derived] Olney DK, Pedehombga A, Ruel MT, Dillon A. A 2-year integrated agriculture and nutrition and health behavior change communication program targeted to women in Burkina Faso reduces anemia, wasting, and diarrhea in children 3-12.9 months of age at baseline: a cluster-randomized controlled trial. J Nutr. 2015 Jun;145(6):1317-24. doi: 10.3945/jn.114.203539. Epub 2015 Apr 22. PMID 25904734